CLINICAL TRIAL: NCT05548985
Title: : Oral Midodrine for Prophylaxis Against Post Spinal Anaesthesia Hypotension During Hip Arthroplasty in Elderly Population: A Randomized Controlled Trial
Brief Title: Midodrine for Prophylaxis Against Post Spinal Hypotension in Elderly Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Hasanin, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MD-25-2021
Record Dates: First submitted 2022-09-17; First posted 2022-09-22 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Hypotension; Spinal Anesthesia; Elderly
MeSH Terms: conditions — Hypotension | interventions — Midodrine; Metoclopramide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Placebo Comparator): oral metoclopramide 10 mg, Metoclopramide tablet was chosen as a placebo because it has the same appearance of midodrine tablet with no cardiovascular effects
  Interventions: Drug: Metoclopramide
- Midodrine group (Active Comparator): oral midodrine tablet (5 mg)
  Interventions: Drug: Midodrine Oral Tablet

INTERVENTIONS:
Drug: Midodrine Oral Tablet — oral midodrine tablet (5 mg) 90 min before performing spinal block
  Arms: Midodrine group
Drug: Metoclopramide — oral placebo (metoclopramide 10 mg tablet). 90 min before performing spinal block
  Arms: control group

SUMMARY:
Hip fracture is a common and serious healthcare problem which commonly affects elderly populations. The common route of anesthesia for hip arthroplasty is spinal anesthesia. Elderly populations are characterized by high incidence of post spinal anesthesia hypotension; furthermore, elderly patients commonly have systemic medical disorder; therefore, this population is highly vulnerable to perioperative hypotension. Moreover , intraoperative hypotension during hip surgery has been recently recognized as a major risk factor for postoperative morbidity and mortality.

Through the effect of spinal anesthesia on sympathetic system Veno-dilatation, decreased venous return, and consequently decreased cardiac output and hypotension will be induced. Vasopressors are commonly used for prophylaxis against post spinal hypotension in different patient subgroups. The commonly used drugs are alpha-adrenoreceptor agonists such as ephedrine, phenylephrine, and recently norepinephrine. All these agents are effective in maintenance of blood pressure; however, they have some disadvantages; ephedrine is commonly associated with tachycardia, phenylephrine and norepinephrine are associated with bradycardia. All the former mentioned drugs are used intravenously.

Midodrine hydrochloride is another alpha-adrenoreceptor agonist drug which is used for management of various hypotensive disorders. Midodrine is the prodrug which is metabolized to desglymidodrine which is a direct arteriolar and venous vasopressor. Midodrine is characterized by being an oral drug, with minimal central nervous system side effects, and good oral bioavailability. No studies had evaluated the efficacy of midodrine for prophylaxis against post-spinal anesthesia hypotension in elderly population.

Aim of the work:

This thesis aims to evaluate the efficacy and safety of oral 5 mg of midodrine compared to placebo in prophylaxis against post-spinal hypotension in elderly patients undergoing hip arthroplasty

DETAILED DESCRIPTION:
Participants will be instructed to fast for 6 hours for solid light meals and 2 hours for clear fluids. The baseline blood pressure will be measured in the preparation room 90 min before spinal anaesthesia as the mean of three measurements with difference of less than 10%. The patients will receive the study drug after measurement of the baseline blood pressure reading. The patient will be monitored for blood pressure and heart rate at 15 min intervals after administration of the study drug. In the operating room, routine monitors (Electrocardiogram, pulse oximetry, and non-invasive blood pressure monitor) will be applied; intravenous line will be secured, and routine pre-medications will be administrated.

Preoperative evaluation of volume status:

All patients will be assessed for volume status before spinal block through evaluation of the inferior vena cava (IVC) collapsibility, and patients who will show IVC collapsibility > 36% will be considered fluid responders and will receive Ringer's lactate solution, 6 mL/kg ideal body weight over 15 minutes.

IVC collapsibility will be calculated as: (maximum IVC diameter - minimum IVC diameter) / maximum IVC diameter.

Anaesthetic management:

Spinal anaesthesia will be performed in the sitting position at level of L3-4 or L4-5 interspaces with a 25-gauge spinal needle. After confirming cerebrospinal fluid flow, 10 mg of 0.5% hyperbaric bupivacaine plus 25 mcg fentanyl will be injected. The degree of sensory block (cold test by alcohol gauze) will be assessed in the study with a goal of T6-8 dermatomal level block. If spinal anaesthesia failed, the patient will be excluded from the study and will be managed according to the attending anaesthetist discretion, local expertise and clinical practice. After induction of spinal anaesthesia maintenance fluid as 2ml/kg/hour of ringer acetate will be commenced.

Post spinal hypotension will be defined as mean arterial pressure < 80% of the baseline reading 30 minutes after spinal block. Hypotension will be managed by 10 mg ephedrine. Severe hypotension will be defined as mean arterial pressure < 70% of the baseline reading and will be managed by 15 mg ephedrine. The dose of ephedrine will be repeated if the hypotensive episode persisted 2 min after the initial bolus. Bradycardia will be defined as heart rate < 50 bpm and will be managed with 0.5 mg of atropine IV.

Blood loss will be replaced using Ringer's lactate solution at a ratio of 3:1 until transfusion threshold is reached. Further blood loss will be replaced using packed RBCs

ELIGIBILITY:
Inclusion Criteria:

* Elderly patients (>65).
* ASA I-II-III.
* Scheduled for hip joint surgery under spinal anaesthesia

Exclusion Criteria:

* • Uncontrolled hypertension

  * Liver cell failure (child B or C).
  * Chronic renal failure on regular dialysis
  * Contraindications of spinal anaesthesia
  * History of allergy to midodrine
  * Cardiac morbidities (impaired contractility with ejection fraction < 50%, heart block, arrhythmias, tight valvular lesions).
  * Acute renal disease, urinary retention
  * Patients on negative chronotropic drugs (such as beta blocker) or vasoconstrictor
  * Patients with glaucoma

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 58 (Actual)
Dates: Start 2022-10-17 (Actual); Primary Completion 2023-07-15 (Actual); Study Completion 2023-07-15 (Actual)

PRIMARY OUTCOMES:
Intraoperative ephedrine consumption | 1 minutes after spinal injection until 45 minutes after induction of spinal anesthesia
  mg

SECONDARY OUTCOMES:
Incidence of post-spinal hypotension | 1 minutes after spinal injection until 45 minutes after induction of spinal anesthesia
  defined as mean arterial pressure < 80% of the baseline reading 45 minutes after induction of spinal anesthesia and not related to blood loss
Incidence of severe spinal induced hypotension | 1 minutes after spinal injection until 45 minutes after induction of spinal anesthesia
  defined as mean arterial pressure < 60% of the baseline reading 45 minutes after induction of spinal anesthesia and not related to blood loss
Incidence of bradycardia | 1 minutes after spinal injection until 45 minutes after induction of spinal anesthesia
  as heart rate less than 50 beats per minutes
heart rate | 1 minute after intervention, every 15 minutes after intervention for 90 minutes, every 2 minutes after spinal anesthesia for 20 min, then every 5 minutes until the end of the procedure
  beats per minutes
mean arterial pressure | 1 minute after intervention, every 15 minutes after intervention for 90 minutes, every 2 minutes after spinal anesthesia for 20 min, then every 5 minutes until the end of the procedure
  mmHg

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
data supporting this research will be available from the PI upon reasonable request

REFERENCES:
- [Derived] Amin S, Hasanin A, Mansour R, Mostafa M, Zakaria D, Arafa AS, Yassin A, Ziada H. Oral midodrine for prophylaxis against post-spinal anesthesia hypotension during hip arthroplasty in elderly population: a randomized controlled trial. BMC Anesthesiol. 2024 Feb 14;24(1):64. doi: 10.1186/s12871-024-02442-8. PMID 38355397